CLINICAL TRIAL: NCT06564402
Title: Augmentation of Exposure Using Positive Mental Rehearsal in Individuals With Increased Social Anxiety
Acronym: APEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Christoph Benke, Principal Investigator, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APEX_SOCIALANX
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Social Anxiety; Social Phobia
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure + Positive Mental Rehearsal (Experimental): Mental rehearsal of the positive aspects of exposure experience
  Interventions: Behavioral: Positive Mental Rehearsal; Behavioral: Exposure
- Exposure + Mental rehearsal (Active Comparator): Mental rehearsal of the exposure experience
  Interventions: Behavioral: Mental Rehearsal; Behavioral: Exposure

INTERVENTIONS:
Behavioral: Positive Mental Rehearsal — After exposure trial, participants are asked about the positive aspects of their exposure experience (e.g., thoughts, feelings), based on which an imagination script is formulated and recounted
  Arms: Exposure + Positive Mental Rehearsal
Behavioral: Mental Rehearsal — After exposure, participants are asked about what happened during the exposure experience and whether their central concerns/expected outcome actually occurred during exposure
  Arms: Exposure + Mental rehearsal
Behavioral: Exposure — All participants complete exposure exercises (i.e., talking on the phone and talking with a stranger) before positive mental rehearsal is executed

SUMMARY:
Efficacy of an optimized exposure therapy training is investigated in individuals with heightened social anxiety. Participants will undergo a one-session standardized exposure training, followed by either standard or positive mental rehearsal of the exposure experience. The efficacy is measured by symptom improvement according to subjective ratings one week later.

DETAILED DESCRIPTION:
Exposure therapy is widely recognized as the gold-standard treatment for anxiety disorders, but its clinically significant response rates remain around 50%. Thus, innovative approaches are needed to improve the efficacy of exposure therapy. One strategy is the mental rehearsal of exposure treatment as a way of supporting the retrieval and consolidation of the exposure memory, which has been demonstrated to be an effective supplement to exposure therapy in a recent study. New conceptualizations also emphasize the role of reward processing and its importance in extinction learning. Several strategies have been proposed to target these reward processes to improve the outcomes of exposure therapy. The present study will examine the use of a positive-focused rehearsal strategy. Participants in the optimized exposure group will engage in an imaginal recounting task focusing on the positive aspects (i.e. emotions, thoughts, behavior) of the exposure. Rehearsal of the positive aspects may increase positive affect, with positive mood thought to be associated with deeper mental rehearsal of stored information. Therefore, the efficacy of using positive mental rehearsal (i.e., imaginal recounting) post-exposure will be investigated, with the use of standard mental rehearsal as an active control group. Participants will be asked to repeat the rehearsal experience at home at two-day intervals. Post-treatment assessment will be conducted one week later. The study will be conducted on healthy participants with an elevated level of social anxiety. The aim of this randomized controlled trial in healthy individuals with increased social anxiety is to investigate whether optimized exposure training (exposure + positive mental rehearsal) is more effective in reducing fear of social interaction compared to an active control group (exposure + mental rehearsal).

ELIGIBILITY:
Inclusion Criteria:

* Elevated score on Social Interactions Anxiety Scale (SIAS) > 26

Exclusion Criteria:

* Current psychotherapeutic/psychiatric treatment
* Plans to start psychotherapeutic/psychiatric treatment in upcoming weeks
* Current suicidal intent
* Severe cardiovascular, respiratory or neurological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Social Interaction Anxiety Scale (SIAS) | Change from baseline to post-treatment (i.e., 7-9 days)
  20-item questionnaire on a 5-point Likert scale (0 = 'not at all'; 4 = 'very strongly') assessing severity of anxiety experienced in social interactions and situations. Total score range: 0 to 80. Higher scores indicate higher severity of social anxiety.
Liebowitz Social Anxiety Scale (LSAS) | Change from baseline to post-treatment (i.e., 7-9 days)
  2-items from the Liebowitz Social Anxiety Scale (LSAS) on a 4-point Likert scale (fear: 0 = 'none'; 3 = 'high'; avoidance: 0 = 'never'; 3 = 'usually') assessing fear and avoidance of the in the intervention exposed situations. Higher scores indicating greater level of fear and avoidance.
Communication Anxiety Inventory (CAI) - Trait Version | Change from baseline to post-treatment (i.e., 7-9 days)
  21-item questionnaire on a 4-point Likert scale (0 = 'almost never'; 3 = 'almost always') assessing an individual's general level of anxiety in communication situations. Total range score: 0 to 84. Higher scores indicate greater level of communication anxiety.

SECONDARY OUTCOMES:
Communication Anxiety Inventory (CAI) - State Version | Baseline
  20-item questionnaire on a 4-point Likert scale (0 = 'not at all'; 3 = 'very strongly' assessing an individual's level of anxiety related to a specific communication situation.
Positive and Negative Affect Schedule (PANAS) | Change from baseline to post-treatment (i.e., 7-9 days)
  20-item questionnaire on a 5-point Likert scale (0 = 'not at all'; 4 = 'extremely' assessing the presence and intensity of both positive and negative emotions. Total score range for positive affect (PA) and negative affect (NA), respectively: 0 to 50. Higher scores indicate on either scale indicate a higher level of that emotion.
Post-Event Processing Inventory (PEPI) - Trait Version | Change from baseline to post-treatment (i.e., 7-9 days)
  12-item questionnaire on a 5-point Likert scale (0 = 'strongly disagree; 4 = 'strongly agree') assessing an individual's general tendency to engage in post-event processing. Total score range: 0 to 60. Higher total scores indicate a greater tendency to ruminate or engage in negative post-event processing.
Post-Event Processing Inventory (PEPI) - State Version | Post-treatment
  12-item questionnaire on a 5-point Likert scale (0 = 'strongly disagree; 4 = 'strongly agree') assessing an individual's level of rumination or post-event processing related to a specific context/situation. Total score range: 0 to 60. Higher total scores indicate a greater engagement in rumination and post-event processing.
Plymouth Sensory Imagery Questionnaire (PSI-Q) | Baseline
  21-item questionnaire across five modalities (visual, auditory, olfactory, gustatory, tactile, and kinesthetic imagery) on a 10-point Likert scale (0 = 'not at all'; 9 = 'mental image as clear and vivid as in real life') assessing how intensively and in detail people can imagine sensory experiences in their mind. Total score range: 0 to 210. Higher total scores indicate a more vivid and detailed sensory imagination.
Snaith-Hamilton-Pleasure-Scale (SHAPS) | Change from baseline to post-treatment (i.e., 7-9 days)
  14-item questionnaire on a 4-point Likert scale (0 = 'strongly disagree'; 3 = 'strongly agree') measuring anhedonia. Scores are transformed to a dichotomous scale: 0 = absence of anhedonia; 1 = presence of anhedonia). Total score range: 0 to 14. Higher total scores indicate greater levels of anhedonia.

CONTACTS AND LOCATIONS:
Locations (1):
- Germany Philipps University, Marburg, Germany

REFERENCES:
- [Background] Rosenberg BM, Barnes-Horowitz NM, Zbozinek TD, Craske MG. Reward processes in extinction learning and applications to exposure therapy. J Anxiety Disord. 2024 Aug;106:102911. doi: 10.1016/j.janxdis.2024.102911. Epub 2024 Jul 29. PMID 39128178
- [Background] McGlade AL, Craske MG. Optimizing exposure: Between-session mental rehearsal as an augmentation strategy. Behav Res Ther. 2021 Apr;139:103827. doi: 10.1016/j.brat.2021.103827. Epub 2021 Feb 11. PMID 33607459
- [Background] Craske MG, Meuret AE, Echiverri-Cohen A, Rosenfield D, Ritz T. Positive affect treatment targets reward sensitivity: A randomized controlled trial. J Consult Clin Psychol. 2023 Jun;91(6):350-366. doi: 10.1037/ccp0000805. Epub 2023 Mar 9. PMID 36892884
- [Background] Craske MG, Meuret AE, Ritz T, Treanor M, Dour H, Rosenfield D. Positive affect treatment for depression and anxiety: A randomized clinical trial for a core feature of anhedonia. J Consult Clin Psychol. 2019 May;87(5):457-471. doi: 10.1037/ccp0000396. PMID 30998048